CLINICAL TRIAL: NCT05404204
Title: Strategy to ROTAblate and PACE (ROTA-PACE) Study
Brief Title: The Efficacy and Safety of a Novel Adjunctive Pacing Strategy During Rotational Atherectomy
Acronym: ROTA-PACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vancouver Island Health Authority (Other)
Responsible Party: Principal Investigator, Bilal Iqbal, Doctor, Vancouver Island Health Authority
Other Study IDs: ROTA-PACE
Record Dates: First submitted 2022-05-26; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease; Coronary Artery Calcification; Bradycardia
Keywords: Coronary Artery Calcification; Rotational Atherectomy; Temporary Pacemaker
MeSH Terms: conditions — Coronary Artery Disease; Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronary artery narrowings interfere with blood flow to the heart which can cause chest pain and heart attacks. Cardiologists can treat these narrowings with balloons and stents. However, some narrowings can become very calcified and hard making treatment with balloons and stents difficult. Rotational atherectomy is a tool to treat calcific coronary disease. It uses an ablative drill to break down the hardened plaques inside the coronary arteries facilitating subsequent treatment with balloons and stents. However, during this procedure patients can experience a slow heart rate which may compromise procedural safety. Cardiologists may use a temporary pacemaker that is inserted by separately accessing the heart through a large vein usually from the leg. This maintains a safe heart rate throughout the procedure. However, inserting the temporary pacemaker is associated with additional complications. We have developed and propose an alternative strategy to provide a temporary safety pacemaker during rotational atherectomy without the need for inserting an additional pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years
* Undergoing percutaneous coronary intervention for angina or acute coronary syndrome.
* Calcific coronary disease requiring rotational atherectomy

Exclusion Criteria:

* Pre-existing pacemaker or implantable cardioverter defibrillator.
* Mobitz II heart block or complete heart block.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing rotational atherectomy for calcific coronary disease without any exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Successful ventricular pacing | At the start of the PCI procedure immediately prior to rotational atherectomy
  Ability to obtain successful ventricular capture prior to rotational atherectomy
Ventricular pacing threshold | At the start of the PCI procedure immediately prior to rotational atherectomy
  The pacing threshold to obtain successful ventricular capture

SECONDARY OUTCOMES:
Complications | At the end of the PCI procedure
  (a) Coronary wire-related intractable spasm (unresponsive to vasodilator therapy); (b) coronary wire-related perforation; (c) New atrial or ventricular arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Iqbal, MD PhD FRCPC, Principal Investigator — Royal Jubilee Hospital, Victoria
Locations (1):
- Royal Jubilee Hospital, Victoria, British Columbia, Canada

REFERENCES:
- [Derived] Iqbal MB, Robinson SD, Nadra IJ, Das D, van Zyl M, Sikkel MB, Della Siega A. The Efficacy and Safety of an Adjunctive Transcoronary Pacing Strategy During Rotational Atherectomy: ROTA-PACE Study. JACC Cardiovasc Interv. 2023 Sep 11;16(17):2189-2190. doi: 10.1016/j.jcin.2023.05.022. Epub 2023 Jul 5. No abstract available. PMID 37409992